CLINICAL TRIAL: NCT01739699
Title: The Efficacy of Intravenous Acetaminophen During The Perioperative Period Of Neurosurgical Patients Undergoing Craniotomies
Brief Title: The Efficacy of Intravenous Acetaminophen During Perioperative Neurosurgery Period
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Endeavor Health (Other)
Collaborators: Cadence Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Steven Greenberg, MD, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EH11-380
Record Dates: First submitted 2012-11-28; First posted 2012-12-03 (Estimated); Results first posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Craniotomy; Brain Surgery
Keywords: craniotomy; brain surgery; acetaminophen; Tylenol
MeSH Terms: interventions — Acetaminophen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetaminophen (Experimental): Subjects will receive 1000mg of intravenous acetaminophen every 6 hours for 24 hours beginning with dural closure.
  Interventions: Drug: Acetaminophen
- Placebo (Other): Subjects will receive 100cc of normal saline every 6 hours for 24 hours beginning at dural closure.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetaminophen
  Other Names: Tylenol
  Arms: Acetaminophen
Drug: Placebo
  Other Names: normal saline
  Arms: Placebo

SUMMARY:
This is a prospective randomized double blinded trial study involving 128 patients undergoing any craniotomy procedure at Evanston Hospital. The patients will be randomized by the sealed envelope technique. The anesthesiologist and nurses who will be administering the placebo or intravenous acetaminophen will be blinded to the group in which patients are assigned.

The following general perioperative data will be recorded: patient information/preoperative data, procedural information, postoperative information, and overall satisfaction of pain management at 24 hours after surgery.

Based on a pilot study (N-20) we expect that 25% of the placebo treated patients will require no opioids in the first 24 hour postoperative period. With the use of intravenous acetaminophen, it is hypothesized that the number of patients that do not require opioids in the first 24 hours after surgery will double.

DETAILED DESCRIPTION:
This is a prospective randomized double blinded trial study involving 128 patients undergoing any craniotomy procedure at Evanston Hospital. The patients will be randomized by the sealed envelope technique. The anesthesiologist and nurses who will be administering the placebo or intravenous acetaminophen will be blinded to the group in which patients are assigned.

The following information will be recorded for each patient enrolled in this study:

* Patient information/Preoperative Data

  * Age, sex, height, weight,
  * Disease specific information
  * Primary diagnosis
  * Pertinent medical history
  * Medications
  * Pertinent changes in patient status
* Procedural information

  * Operation type
  * Preoperative anesthetic medications
  * Induction meds, intra-operative anesthetic meds, and post-operative anesthetic meds
  * Duration of Surgery and Intubation
  * Amount of dilaudid equivalent narcotics
* Postoperative Information

  * Amount of narcotics administered in the PACU
  * Amount of narcotics administered in the first 24 hour postoperative period
  * Amount of non-narcotic analgesics administered in the first 24 hour postoperative period
  * Time to first rescue analgesic in the PACU
  * Amount of first rescue medication recorded
  * Assessment of Pain Intensity at T0.5 (30min into PACU stay) and T24 (24 hours after end of surgery) (A 10-cm VAS scale will be used and labeled no pain at its left terminus and worst pain imaginable at its right terminus)
  * Temperature in degrees centigrade every 8 hours for 24hours.
  * CAM-ICU is performed by ICU nurses to detect delirium in patients every 8 hours and will be documented on a data collection sheet for the first 24 hours
  * RASS is a sedation scoring system that is used in our ICU and is documented every 8 hours by ICU nursing. We will record the RASS score for the first 24 hours on a data collection sheet as documented by the ICU nurse.
  * Overall satisfaction score at 24 hrs. "Overall satisfaction with pain management" (verbal rating score: scale 1 - 100)

Based on a pilot study (N-20) we expect that 25% of the placebo treated patients will require no opioids in the first 24 hour postoperative period. With the use of intravenous acetaminophen, it is hypothesized that the number of patients that do not require opioids in the first 24 hours after surgery will double.

ELIGIBILITY:
Inclusion Criteria:

* Subject are able to provide informed consent prior to participation in the study
* Subjects must be scheduled to undergo elective open craniotomy procedure of > 2 hour duration
* Subjects must be >18 years old but less than 90 years old
* Subjects must have an American Society of Anesthesiologists (ASA) class I-IV
* Subjects must have the ability to communicate meaningfully with the investigator staff and read/understand the study procedures and the use of pain scales

Exclusion Criteria:

* Subjects used opioids or tramadol daily for >7 days before study medication administration
* Subjects had been treated with any of the following within 14 days of surgery: chaparral, comfrey, germander, jin bu huan, kava, pennyroyal, skullcap, St. John's wort, or valerian
* Subjects who have a chronic pain condition, significant medical disease or laboratory abnormality that in the investigator's judgment could compromise the subject's welfare
* Subjects with known hypersensitivity to opioids, acetaminophen or the inactive ingredients
* Subjects with known or suspected history of alcohol or drug abuse or dependence in the previous 2 years prior to the proposed surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2012-01; Primary Completion 2016-08-01 (Actual); Study Completion 2017-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Greenberg, MD, Principal Investigator — NorthShore University Health Sytem - Evanston Hospital Department of Anesthesia
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Data is stored in file at our system
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: anytime
Access Criteria: anytime

RESULTS

PARTICIPANT FLOW:
Groups:
- Acetaminophen: Subjects will receive 1000mg of intravenous acetaminophen every 6 hours for 24 hours beginning with dural closure.
  Acetaminophen
- Placebo: Subjects will receive 100cc of normal saline every 6 hours for 24 hours beginning at dural closure.
  Placebo
Period: Overall Study
Arm/Group | Acetaminophen | Placebo
Started | 70 | 70
Completed | 66 | 65
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetaminophen | Placebo | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 45 | 91
  >=65 years | 24 | 25 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (15) | 56 (13) | 57 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 36 | 77
  Male | 29 | 34 | 63
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 70 | 70 | 140

OUTCOME MEASURES:

1. Primary Outcome: Opioid Requirement After Surgery
Description: The purpose of the study was to determine whether more patients undergoing craniotomies would not require any opioids (i.e., opioid consumption reduced to zero) during the first 24 postoperative hours when receiving intravenous (IV) acetaminophen during that time compared to those receiving placebo (normal saline).
Time Frame: during first 24 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 66 | 65
Participants | 10 | 4

2. Secondary Outcome: Time to Rescue Medication in Both Groups
Description: Time (minutes) from end of procedure to first rescue dose in either PACU or ICU
Time Frame: 0 to 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 66 | 65
minutes | 22 [16.5 to 33] | 37 [20.5 to 53.5]

3. Secondary Outcome: Amount of Rescue Medication in PACU in Both Groups
Time Frame: 0 to 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 66 | 65
mg | 0.5 [0.3 to 0.5] | 0.5 [0.3 to 0.5]

4. Secondary Outcome: Median Difference in ICU Length of Stay/Hospital Length of Stay Between Both Groups
Time Frame: from 0 to estimated 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 66 | 65
hours
  Hospital Length of stay | 71.75 [49 to 118] | 75.5 [50 to 119]
  ICU length of stay | 26 [21.5 to 41] | 28 [22 to 52.5]

5. Secondary Outcome: Number of Participants Who Had a Successful Neurologic Exams Between Intervention and Placebo Group as Determined by a Neurosurgical Provider by Answering Either Yes or No
Description: Successful neurologic exams are performed by neurosurgical team during the first 24 hour period. Successful neurologic exams will be provided by a neurosurgical professional and they will answer Yes or No if the exam is appropriate.
Time Frame: from 0 to estimated maximum of 24 hours after surgery
Population: As length of stay increased in ICU, the likelihood of discharge increased for the patients. This lowered the total amount of analyzed patients as the time increased.
Measure: Count of Participants; unit: Participants
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 66 | 65
Participants
  ICU arrival: number analyzed (Participants) | 64 | 65
  ICU arrival | 57 | 61
  8 Hours: number analyzed (Participants) | 64 | 65
  8 Hours | 63 | 64
  16 Hours: number analyzed (Participants) | 63 | 62
  16 Hours | 60 | 60
  24 Hours: number analyzed (Participants) | 58 | 58
  24 Hours | 53 | 55

6. Secondary Outcome: Median Difference in Temperature Between Intervention and Placebo Groups
Description: Temperature measure in degrees celcius during the first 24hours postoperatively in increments of 8 hours.
Time Frame: from 0 to estimated maximum 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: Degrees Celcius
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 66 | 65
Degrees Celcius
  ICU Arrival | 36.6 [36.4 to 36.8] | 36.7 [36.4 to 36.8]
  8 Hours | 36.7 [36.5 to 36.9] | 36.8 [36.6 to 37.0]
  16 Hours | 36.7 [36.5 to 37.0] | 36.8 [36.6 to 37.0]
  24 Hours | 36.8 [36.6 to 37.0] | 36.7 [36.5 to 37.0]

7. Secondary Outcome: Sedation Scores Measured by Richmand-Agitation-Sedation Scale (RASS) Every 8 Hours for 24 Hours in Both Groups
Description: Sedation scores will be evaluated by providers through the Richmand-Agitation-Sedation Scale (RASS) system every 8 hours for the first 24hour postoperatively. The RASS is a 10 point scale with four levels for anxiety or agitation (+1 to +4 (indicates more agitation and alertness the higher number you have)), one level to indicate a calm and alert state (0), and 5 levels of deeper sedation (-1 to -5 ( the more negative number indicating a deeper level of sedation)) patients. It helps guide sedation therapy at the bedside. There are no worse outcomes with different levels of sedation scores. However, typically, we try to keep the scores in the range of 0-+1 to be able to appropriately assess patients and allow them to be mobile in a safe fashion.
Time Frame: during first 24 hours after surgery
Population: The amount of participants analyzed decreased as length of stay in the ICU increased as patients were likely discharged from the ICU. The median number indicates the RASS score and not the number of participants.
Measure: Median (Inter-Quartile Range); unit: median of RASS scores
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 66 | 65
median of RASS scores
  ICU arrival | 0 [-1 to 0] | 0 [-1 to 0]
  8 hours: number analyzed (Participants) | 63 | 64
  8 hours | 0 [0 to 0] | 0 [0 to 0]
  16 hours: number analyzed (Participants) | 62 | 63
  16 hours | 0 [0 to 0] | 0 [0 to 0]
  24 hours: number analyzed (Participants) | 57 | 57
  24 hours | 0 [0 to 0] | 0 [0 to 0]

8. Secondary Outcome: Pain VAS Scores (1-100) Every 8 Hours for 24 Hours in Both Groups
Description: Pain was measured using the Visual Analog Scale (VAS) for each patient at the time of arrival and every eight hours after arrival for the first 24 hours of ICU stay. A VAS score of 1 indicates little or no pain and a VAS score of 100 indicates severe pain.
Time Frame: during first 24 hours after surgery
Population: The median number below indicates the median VAS score.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 66 | 65
units on a scale
  ICU Arrival | 35 [20 to 60] | 50 [10 to 70]
  8 Hours | 30 [10 to 50] | 45 [20 to 60]
  16 Hours | 30 [10 to 50] | 30 [10 to 60]
  24 Hours | 30 [10 to 50] | 20 [10 to 50]

9. Secondary Outcome: # of Participants With Delirium Measured by a Positive CAM-ICU Every 8 Hours for 24 Hours in Both Groups-
Description: Delirium was assessed in each of the participants upon arrival to the ICU using the Confusion Assessment Method for the ICU (CAM-ICU). The CAM-ICU was performed for each participant every 8 hours following admission for the first 24 hours
  The CAM ICU scoring is based on a scale of 0-7, 0-2=no delirium, 3-5=miild delirium, 6-7=severe delirium. The positive CAM ICU consists of features 1 and 2 and either 3 or 4:
  Features 1: Acute onset or fluctuating course Features 2: Inattention Features 3: Disorganized thinking Features 4: Altered level of consciousness
Time Frame: during first 24 hours after surgery
Population: As the time post surgery increased, the amount of individual participants discharged from the ICU increased.
Measure: Count of Participants; unit: Participants
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 66 | 65
Participants
  ICU Arrival: number analyzed (Participants) | 64 | 65
  ICU Arrival | 1 | 0
  8 Hours: number analyzed (Participants) | 65 | 65
  8 Hours | 0 | 0
  16 Hours: number analyzed (Participants) | 64 | 64
  16 Hours | 0 | 0
  24 Hours: number analyzed (Participants) | 59 | 57
  24 Hours | 0 | 0

10. Secondary Outcome: Median Satisfaction Scores on a Verbal Score From 1(Not Satisfied at All) to 100 (Very Satisfied)
Description: on a verbal score 1-100, 1 would mean that the patient is not satisfied at all and 100 would mean that the patient was very satisfied.
Time Frame: During first 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 66 | 65
units on a scale | 87.5 [55 to 100] | 80 [50 to 100]

ADVERSE EVENTS:
Time Frame: Any adverse events were noted for 7 days following completion of the procedure.
Arm/Group | Acetaminophen | Placebo
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/65
Other Adverse Events (participants affected / at risk) | 0/66 | 0/65

LIMITATIONS AND CAVEATS:
1. Underpowered.
2. Nurses used the local standard order sets.
3. Dexamethasone dose was not standardized
4. Long acting opioids or NSAIDS of any type were not administered.
5. Patients observed every 8 hours for 24 hours postoperatively.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No